CLINICAL TRIAL: NCT06406959
Title: The Effect of Preemptive Regional Anesthesia (TAP-block) on Acute and Chronic Pain After Transabdominal Preperitoneal Inguinal Hernia Repair (TAPP) - a Randomized Controlled Trial
Brief Title: The Effect of Preemptive Regional Anesthesia (TAP-block) on Acute and Chronic Pain After Transabdominal Preperitoneal Inguinal Hernia Repair (TAPP)
Acronym: ERA-TAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Taras V. Nechay, MD, Professor, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2024-04-20; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Primary Inguinal Hernia
Keywords: transverse abdominis plane block; inguinal hernia; TAPP technique; chronic postoperative pain; acute pain; inguinal hernia surgery
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP-block (Experimental): TAPP inguinal hernia repair under general anesthesia with endotracheal intubation. Patients receive unilateral US-guided TAP-block with 20 ml 0,375% Levobupivacaine before incision
  Interventions: Procedure: Transversus abdominal plane block (TAP block)
- Standard care (No Intervention): TAPP inguinal hernia repair under general anesthesia with endotracheal intubation (without preemptive regional anesthesia) in accordance with actual standard of care.

INTERVENTIONS:
Procedure: Transversus abdominal plane block (TAP block) — Unilateral US-guided TAP-block lateral approach with 20 ml 0,375% Levobupivacaine before incision
  Arms: TAP-block

SUMMARY:
The study is devoted to the impact of preemptive regional Transversus abdominal plane block on the postoperative acute and chronic pain after elective Transabdominal preperitoneal (TAPP) inguinal hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most common elective interventions in general surgery. Approximately 20 million inguinal hernia repairs are performed worldwide every year. Laparo-endoscopic techniques provide faster recovery times, lower chronic pain risk and are cost effective compared to open one.

Nevertheless, laparoscopic inguinal hernia repair can result in moderate to severe pain in the early postoperative period, interfering the time of returning to normal activity in a substantial quantity of patients. To reduce pain and to accelerate recovery, local and regional anesthetics has been successfully implemented into the daily routine of abdominal surgeries.

Recent systematic reviews have shown that TAP block can reduce analgetic consumption and acute pain scores after inguinal hernia repair. However, most included studies were conducted on patients with open hernia surgery or total extra peritoneal (TEP) inguinal hernia repair. Some studies showed the benefit of TAP block for early pain control following TAPP. Most of them were retrospective, some conducted with exclusion of obese or comorbid patients, some in mixed groups without separating patients with TAPP and TEP.

Thus, the evidence of TAP block efficiency prior to hernia repair in TAPP technique are of low quality.

Chronic postoperative inguinal pain (CPIP) develops in up to 6% of patients after TAPP. Several studies have found that intense acute postoperative pain is a risk factor for CPIP after IHR. The investigators hypothesize, that preemptive TAP block temporary stops nociception and central sensitization from the surgical site thus reduce acute postoperative pain that theoretically provoke reducing the incidence of CPIP following IHR. Two studies suggest that TAP block may influence the incidence of CPIP after TAPP. Considering the retrospective study design of both and the insufficient sample size further randomized clinical trials are mandatory to estimate this hypothesis.

The aim of our study is to explore the possibilities of reducing acute and chronic pain after TAPP via implementation TAP block.

The sample size was calculated based on the randomized controlled trial data of patients after TEP IHR where postoperative VAS score at 4 h on coughing was 4.7±1.5 in the preemptive local anesthesia group and 6.1±1.9 in the control group. A sample size of 39 patients was required for each subgroup (total=78 patients) with a type I error rate α=0.05 and type II error rate β=0.1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral primary inguinal hernia who are scheduled for elective Transabdominal preperitoneal inguinal hernia repair (TAPP)
* Signed Informed consent to participation
* ASA I-III
* BMI ≤35 kg/m2

Non-inclusion Criteria:

* Inguinoscrotal hernia (hernia passing through the entrance to the scrotum)
* Previously diagnosed mental disorders
* Patients receiving psychotropic drugs and drugs affecting adrenal cortex function (estrogens and systemic glucocorticoids)
* Language barrier

Exclusion Criteria:

* Deviations during the operation/anesthesia that required transfer to the intensive care unit or conversion to open surgery
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain 4h | 4±1 hours postop
  Pain score will be assessed using the Numeric Pain Rating Scale (NRS) (0-10) at rest and on coughing.

SECONDARY OUTCOMES:
Acute postoperative pain 2h | 2±1 hours postop
  Pain score will be assessed using the Numeric Pain Rating Scale (NRS) (0-10) at rest and on coughing.
Acute postoperative pain 6h | 6±1 hours postop
  Pain score will be assessed using the Numeric Pain Rating Scale (NRS) (0-10) at rest and on coughing.
Number of Participants meeting discharge criteria | 6±1 hours postop
  Blood pressure ≥100/60 mm Hg; Activation within the department; Ability to oral medication (no postoperative nausea and vomiting); Pain (NRS) ≤3 points; No signs of complications (bleeding, early relapse)
Analgetic consumption (dose quantity) | 24 hours postop
  At NRS score 4-6 at rest patients receive: 30mg Ketorolak IV no more than once every 8 hours or 1000mg Acetaminophen IV no more than once every 6 hours; At NRS score ≥7 at rest patients receive 100 mg Tramadol IV no more than once every 12 hours; The number of analgesic doses administered is counted.
Concentration of serum cortisol | At 8 am on the day of surgery, 4±1 hours postop
  nmol/L
Acute postoperative pain 24h | 24±3 hours postop
  Pain score will be assessed using the Numeric Pain Rating Scale (NRS) (0-10) at rest and on coughing.
  Participants verbally requested to rate their pain: "Rate your pain from 0 (no pain) to 10 (unbearable pain)". 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Length of stay | From date of hospitalization until the date of discharge
  Days
Number of Participants with postoperative complications | Postoperative 30 (±3) days
  Number of Participants with postoperative complications, evaluated by Clavien-Dindo classification (telephone survey)
Patient satisfaction score | Postoperative 30 (±3) days
  Patient satisfaction with treatment is assessed by telephone survey using the Linkert-type scale (1 - less satisfaction, 5 - more satisfaction)
Number of Participants with chronic pain | Postoperative 90 (±3) days
  Pain score will be assessed by NRS (telephone survey). Participants verbally requested to rate their pain: "Rate your pain from 0 (no pain) to 10 (unbearable pain)". 0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Number of Participants with recurrence | After 90 days
  Participants undergo a telephone survey. Participants presenting with characteristic complaints are invited for examination and ultrasound scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of faculty surgery №1 Pirogov Russian National Research Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aasvang EK, Gmaehle E, Hansen JB, Gmaehle B, Forman JL, Schwarz J, Bittner R, Kehlet H. Predictive risk factors for persistent postherniotomy pain. Anesthesiology. 2010 Apr;112(4):957-69. doi: 10.1097/ALN.0b013e3181d31ff8. PMID 20234307
- [Background] Arora S, Chhabra A, Subramaniam R, Arora MK, Misra MC, Bansal VK. Transversus abdominis plane block for laparoscopic inguinal hernia repair: a randomized trial. J Clin Anesth. 2016 Sep;33:357-64. doi: 10.1016/j.jclinane.2016.04.047. Epub 2016 May 28. PMID 27555193
- [Background] Chamzin A, Frountzas M, Gkiokas G, Kouskouni E, Xanthos T, Michalopoulos NV. The Effect of Intraoperative Transversus Abdominis Plane Blocking on Postoperative Pain After Laparoscopic Transabdominal Pre-peritoneal (TAPP) Groin Hernia Repair. Front Surg. 2022 Feb 8;9:834050. doi: 10.3389/fsurg.2022.834050. eCollection 2022. PMID 35211504
- [Background] Gao T, Zhang JJ, Xi FC, Shi JL, Lu Y, Tan SJ, Yu WK. Evaluation of Transversus Abdominis Plane (TAP) Block in Hernia Surgery: A Meta-analysis. Clin J Pain. 2017 Apr;33(4):369-375. doi: 10.1097/AJP.0000000000000412. PMID 27518492
- [Background] Hosni M, Soulios, JP, Francart, D. Ultrasound transversus abdominis plane (TAP) block versus local infiltration analgesia for acute and chronic postoperative pain control after laparoscopic bilateral hernia repair: a single-center randomized controlled trial. Acta Anaesthesiologica Belgica. 2020; 71(4), 171-174. https://doi.org/10.56126/71.4.2
- [Background] Hubbard G, Hubert C, Vudayagiri L, Tullington J, Merino K, Vaidya A, Gemma R. Transversus abdominis plane blocks in laparoscopic inguinal hernia repair: a review. Hernia. 2023 Oct;27(5):1059-1065. doi: 10.1007/s10029-023-02831-x. Epub 2023 Jul 3. PMID 37395916
- [Background] HerniaSurge Group. International guidelines for groin hernia management. Hernia. 2018 Feb;22(1):1-165. doi: 10.1007/s10029-017-1668-x. Epub 2018 Jan 12. PMID 29330835
- [Background] Kim MG, Kim SI, Ok SY, Kim SH, Lee SJ, Park SY, Lee SM, Jung BI. The analgesic effect of ultrasound-guided transverse abdominis plane block after laparoscopic totally extraperitoneal hernia repair. Korean J Anesthesiol. 2012 Sep;63(3):227-32. doi: 10.4097/kjae.2012.63.3.227. Epub 2012 Sep 14. PMID 23060979
- [Background] Paasch C, Fiebelkorn J, Berndt N, De Santo G, Aljedani N, Ortiz P, Gauger U, Boettge K, Anders S, Full H, Strik MW. The transversus abdominis plane block reduces the cumulative need of analgesic medication following inguinal hernia repair in TAPP technique: a retrospective single center analysis among 838 patients. Hernia. 2020 Dec;24(6):1371-1378. doi: 10.1007/s10029-020-02156-z. Epub 2020 Mar 13. PMID 32170456
- [Background] Paasch C, Fiebelkorn J, De Santo G, Azarhoush S, Boettge K, Anders S, Gauger U, Strik M. The transversus abdominis plane block may reduce chronic postoperative pain one year after TAPP ingunial hernia repair. Ann Med Surg (Lond). 2020 May 23;55:190-194. doi: 10.1016/j.amsu.2020.04.011. eCollection 2020 Jul. PMID 32518639
- [Background] Reinpold W. Risk factors of chronic pain after inguinal hernia repair: a systematic review. Innov Surg Sci. 2017 May 12;2(2):61-68. doi: 10.1515/iss-2017-0017. eCollection 2017 Jun. PMID 31579738
- [Background] Takebayashi K, Matsumura M, Kawai Y, Hoashi T, Katsura N, Fukuda S, Shimizu K, Inada T, Sato M. Efficacy of transversus abdominis plane block and rectus sheath block in laparoscopic inguinal hernia surgery. Int Surg. 2015 Apr;100(4):666-71. doi: 10.9738/INTSURG-D-14-00193.1. PMID 25875548